CLINICAL TRIAL: NCT00238901
Title: Efficacy and Safety of Basiliximab in HCV+ Patients Undergoing Liver Transplantation, as Compared With Steroids, Both Given in Combination With Cyclosporine and Mycophenolate Mofetil (MMF)
Brief Title: Efficacy and Safety of Basiliximab in Hepatitis C Virus Positive Patients Undergoing Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCHI621AIT06
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Liver Transplant
Keywords: Liver transplant, HCV+, steroid free
MeSH Terms: conditions — Hepatitis C | interventions — Basiliximab

INTERVENTIONS:
Drug: Basiliximab

SUMMARY:
The natural history of HCV infection in liver transplant recipients may be accelerated when compared to that in patients with normal immune systems.

The objective of this trial is to assess the efficacy and safety of basiliximab, in combination with cyclosporin and MMF on the success rate of liver transplants for HCV related cirrhosis, in comparison with standard steroid treatment.

ELIGIBILITY:
Inclusion Criteria Patients undergoing first cadaver liver transplant Patients receiving an AB0 identical or compatible graft HCV+ patients (serology test within the last 12 months)

Exclusion Criteria Antiretroviral prophylactic treatment post-transplant Serological markers positive for Hepatitis B surface Antigen and Human Immunodeficiency Virus Recipients of a split liver transplant Other protocol-defined inclusion/exclusion criteria applied

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2002-12; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
12-month cumulative incidence of post-surgical graft loss and death

SECONDARY OUTCOMES:
hepatitis C recurrence (see definition 3.5.2) at 6 and 12 months after transplant surgery.
treated and biopsy proven acute rejection at 6 and 12 months after transplant surgery.
graft survival and patient survival after treatment with either Simulect or steroids at 6 and 12 months.
viral load (HCV-RNA) after treatment with Simulect or steroids at Baseline, Month 1 and 3 post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis